CLINICAL TRIAL: NCT04137679
Title: Efficacy and Safety of Neo-Radiochemotherapy Followed Surgery Compared With Definitive Radiochemotherapy in Patients With Initial Unresectable Esophageal Cancer
Brief Title: Efficacy and Safety of Neo-CRT Followed Surgery Compared With Definitive CRT in Patients With Initial Unresectable ESO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJESO-1
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-08

CONDITIONS: Unresectable Esophageal Cancer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Definitive Radiochemotherapy (Experimental): Concurrent Radiochemotherapy:
  Radiotherapy,IMRT, 60Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day.
  Interventions: Radiation: Definitive Radiochemotherapy; Procedure: Neoadjuvant Radiochemotherapy followed by surgery
- Neoadjuvant Radiochemotherapy followed by surgery (Active Comparator): Concurrent Radiochemotherapy:
  Radiotherapy,IMRT, 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day; Receive radical surgery 4 to 6 weeks later.
  Interventions: Radiation: Definitive Radiochemotherapy; Procedure: Neoadjuvant Radiochemotherapy followed by surgery

INTERVENTIONS:
Radiation: Definitive Radiochemotherapy — Radiotherapy,IMRT, 60Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day
Procedure: Neoadjuvant Radiochemotherapy followed by surgery — Concurrent Radiochemotherapy: Radiotherapy,IMRT, 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day; Receive radical surgery 4 to 6 weeks later.

SUMMARY:
Definitive chemoradiotherapy(CRT) has been regarded as a standard of care for patients with unresectable locally advanced esophageal cancer. Patients who are sensitive to CRT can achieve significantly down staging. Whether this part of patients could benefit from further surgical treatment remains unknown. Herein, a single center prospective randomized phase II clinical trial will be carried out to compare efficacy and safety of definitive CRT versus neo-CRT plus radical resection in patients who achieved down staging after neo-CRT for stage T4NxM0 esophageal Cancer.

DETAILED DESCRIPTION:
1. Compare progression-free survival (PFS) and overall survival (OS) of definitive radiochemotherapy versus(VS) neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who down stage from inoperable to operable after neoadjuvant treatment;
2. Compare the toxic and side effects of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete remission after neoadjuvant treatment;
3. Assess impact of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection on quality of life of patients.

Concurrent Radiochemotherapy: Radiotherapy, Intensity Modulation Radiation Therapy(IMRT), 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2), 1st/8th/15th/22nd day

ELIGIBILITY:
Inclusion Criteria:

1. Thoracic esophageal cancer patients or esophagogastric junction cancer patients, with locally advanced unresectable tumor, clinically identified before treatment as T4bNxM0 or lymph node metastases (LNM)invading adjacent structures according to UICC(International Union Against Cancer) TNM(primary tumor, regional nodes, metastasis) Classification of Malignant Tumours, 8th ed.
2. Initial unresectable assessed by surgeon.
3. Patients able to tolerate surgery.
4. Untreated patients who have not received any antitumor therapy.
5. Life expectancy > 6 months.
6. Age: 18-70 years.
7. White blood cell count ≥4.0×10^9/L, ANC(absolute neutrophil count) ≥1.5×10^9/L, thrombocyte count ≥100×10^9/L, hemoglobin ≥90 g/L; normal liver and kidney functions.
8. WHO PS(Performance Status): 0-1.
9. Patients who understood the study and gave signed informed consent.

Exclusion Criteria:

1. Patients who have already received antitumor therapy, including chemotherapy, radiotherapy or surgery.
2. Patients with hemorrhage or complicated hemorrhage.
3. Other uncontrollable patients who are not suitable for surgery.
4. Patients who deny to accept surgery.
5. Pregnant or lactating women.
6. Patients who agree without acknowledgement as a result of psychological, family or social factors.
7. Patients with CTCAE(Common Terminology Criteria Adverse Events Version 4.0) grade ≥2 peripheral neuropathy.
8. Patients who have ever had malignant tumors other than esophageal cancer.
9. Patients with a history of diabetes for >10 years with unsatisfactory control of blood glucose level.
10. Patients with serious heart, lung, liver or kidney dysfunction, hematopathy, immune system disease or cachexia who therefore cannot tolerate chemotherapy or surgery.
11. Patients with severe infection.
12. Patients with uncontrolled diabetes, random blood glucose > 200mg/L, fasting glucose >140mg/L.
13. Patients with other severe disease, such as myocardial infarction in the last 6 months.
14. Patients who participate in other clinical trials right now or in the last 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Compare overall survival of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant radiochemotherapy
Disease-free survival | 3 years
  Compare progression-free survival of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant radiochemotherapy.

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 5 years
  grade 3 or 4 toxicity of leukocytes, febrile neutropenia, thrombocytes, hemoglobin, nausea/vomiting, diarrhea, stomatitis, esophagitis, cardiovascular.

CONTACTS AND LOCATIONS:
Overall Officials: Qingsong Pang, Doctor, Study Chair — Department of Radiation Oncology, Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No